CLINICAL TRIAL: NCT06492473
Title: Clinical Evaluation Of Ventricular Septal Defect (VSD) in Children at Sohag University Hospital
Brief Title: Clinical Evaluation Of Ventricular Septal Defect (VSD) In Children at Sohag Univesity Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amany Sabry Thabet, Resident of pediatric and neonatology department, Sohag University Hospitals, Sohag University
Other Study IDs: soh-med-24-6-16MS
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Ventricular Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Ventricular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ECHO — type and size of ventricular septal defect

SUMMARY:
ventricular septal defect(VSD) are one of the most common significant CHD and account for up to 40% of all cardiac abnormalities.VSD is commonly isolated defect as well as intrinsic component of several complex cardiac malformations including tetrology of fallot ,double- outlet right ventricle(RV),transposition of great vessles,aortic coartication or interruption ,and truncus arteriosus

ELIGIBILITY:
Inclusion Criteria:

* all children from date of birth to age of 16 years old including both genders diagnosed to have isolated VSD or apart from another cardiac anomalies

Exclusion Criteria:

-

Ages: 1 Day to 16 Years | Sex: All
Age Groups: Child
Study Population: all children from date of birth to age of 16 years old including both genders diagnosed to have isolated VSD or apart from another cardiac anomalies
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-06-24 (Estimated); Study Completion 2025-06-24 (Estimated)

PRIMARY OUTCOMES:
size of VSD | 12 months
  size of VSD in mm according echocardiology

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saxena A, Mehta A, Sharma M, Salhan S, Kalaivani M, Ramakrishnan S, Juneja R. Birth prevalence of congenital heart disease: A cross-sectional observational study from North India. Ann Pediatr Cardiol. 2016 Sep-Dec;9(3):205-9. doi: 10.4103/0974-2069.189122. PMID 27625516
- [Background] Soto B, Becker AE, Moulaert AJ, Lie JT, Anderson RH. Classification of ventricular septal defects. Br Heart J. 1980 Mar;43(3):332-43. doi: 10.1136/hrt.43.3.332. PMID 7437181
- [Background] Soto B, Ceballos R, Kirklin JW. Ventricular septal defects: a surgical viewpoint. J Am Coll Cardiol. 1989 Nov 1;14(5):1291-7. doi: 10.1016/0735-1097(89)90430-0. PMID 2808985
- [Background] Kirklin JK, Castaneda AR, Keane JF, Fellows KE, Norwood WI. Surgical management of multiple ventricular septal defects. J Thorac Cardiovasc Surg. 1980 Oct;80(4):485-93. PMID 7421283